CLINICAL TRIAL: NCT05529602
Title: Comparison of Post Isometric Relaxation and Core Stability Exercises on Pain and Disability in Postpartum Females With Sacroiliac Joint Dysfunction
Brief Title: Post Isometric Relaxation and Core Stability Exercises in Sacroiliac Joint Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0508
Record Dates: First submitted 2022-07-24; First posted 2022-09-07 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Lower Back Pain
Keywords: core stability; Core strengthening; chronic low back pain; therapeutic exercises
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- post isometric relaxation exercises and core stability (Experimental): for pain and disability secondary to SIJ dysfunction in postpartum females
  Interventions: Other: conventional physical therapy
- conventional physical therapy (Other): for management of lower back pain
  Interventions: Other: relaxation exercise

INTERVENTIONS:
Other: conventional physical therapy — core stability exercises
  A total of 3 sessions per week were given for 15-20 minutes
  Arms: post isometric relaxation exercises and core stability
Other: relaxation exercise — the experimental group was given Post-isometric relaxation exercise along with core stability
  A total of 3 sessions per week were given for 15-20 minutes
  Arms: conventional physical therapy

SUMMARY:
There is growing evidence on the effects of post isometric relaxation exercises and core stability exercises on pain and disability secondary to various disorders. However, very few studies have explored their effects in postpartum Sacroiliac joint dysfunction. The aim of this study will be to compare the effects of post isometric relaxation exercises and core stability exercises on pain in postpartum Sacroiliac joint dysfunction.

DETAILED DESCRIPTION:
A previous study conducted by Farhadi et al. assessed that the prevalence of sacroiliac joint pain has been reported between 13-30% in postpartum females aged between 40-and 45 years. Specifically, 13% of the individuals with low back pain have the origin of their pain from the sacroiliac joint. It has been found that 33.6% of pregnant women have pelvic girdle pain, and 18.9% of post-partum women have "serious" pelvic girdle pain. In most women with pregnancy-related sacroiliac, joint pain resolves with time after pregnancy, but in some females, the pain lingers on. Patients with Sacroiliac dysfunction generally complain of pain in their back, and buttock or may radiate to the knee. On examination, there is pain and local tenderness. The symptoms increase on position change such as getting up from a sitting or lying position or while ascending and descending stairs. Sacroiliac pain is localized to the posterior pelvis and is described as stabbing pain deep.

Terzi and Clinton et al., (2019) found thirty women diagnosed with post-partum SIJ pain, their age ranged from (25-35)years, their BMI ranged from (25-to 30)kg/m², and their number of parity ranged(from 2-to 4)times were selected randomly from the outpatient clinic of Al-Ahrar teaching hospital. Women were divided randomly into two equal groups, Group A (Control group): 15 patients, they were treated by TENS for 4 weeks 30 min\session, 3 sessions \week. Group B(Study group):15 patient, were treated with core stability exercises for 4 weeks, 30 min\session, 5 sessions \week plus TENS as for group A. All participant was evaluated by VAS, Oswestry disability index (ODI), serum cortisol levels before and after treatment. The results revealed that there was a statistically significant decrease in the mean value of VAS in the group (B) when compared with its corresponding value in group (A). In spite of there being no statistically significant difference in plasma cortisol level, there was a clinical difference and high percent of improvement in favor of group B (8.83%) over group A (2.66%). Also, there was a statistically significant decrease in the mean value of ODI in the group (B) when compared with its corresponding value in group (A). It was concluded that core stability exercises could be used as a complementary treatment in reducing post-partum SIJ pain. Also, it could be considered a useful treatment to increase flexibility and range of motion.

Shamsi et al., in 2014, found that reduced pain and increased function are outcomes when core stability exercises are used in the early stages of interventions. Also, Huxel et al., found that core exercises resulted in better outcomes measures than general exercise in the first 3 months of interventions for LBP, as they found clinical improvements in pain perception and functional disability levels when the patients with LBP engaged in core-specific exercise.

One study was done by Noelle M.Selkow et al., (2017) supports the findings of our study by concluding that MET is effective in decreasing pain in patients with acute low back pain. Another study was done by Roberts BL where he described two techniques of soft tissue manipulation viz neuromuscular technique and MET and found that MET can reduce Pain, muscle rigidity, and lengthen muscle fibers. The effect of MET on disability is supported by Fenech et al., (2015) determined that LBP is one of the most common musculoskeletal problems that affects about 60-80% of the population throughout their life expectancy. The lifetime prevalence of low back pain is reported to be 84% with 11-12% of the population being disabled by this condition. In 2010 Global Burden of Disease conducted a study on low back pain and estimated the global age-standardized point prevalence to be 9.4%. Low back pain is a self-limiting condition that can commonly be found in middle age ranging from 35 to 65 years and 90% of the people can be cured within 3-4 months without any treatment protocol.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum females with sacroiliac joint dysfunction
* Diagnosed Patients with SIJ dysfunction
* Females who will be physically active
* Age between 20 to 35 years
* Females having a post-partum period

Exclusion Criteria:

* Post Spinal surgery/instrumentation
* prolonged steroid use and bone tissue infection or malignancy)
* Radiculopathy
* Acute Traumatic injury of spine/lower extremity
* Patient under anticoagulant therapy
* Delivery with any complication
* Females have any history of diabetes, hypertension, or any chronic illness
* Any Pelvic or abdominal surgery in past
* Disc herniation or spine fracture

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 54 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
MODIFIED OSWESTRY DISABILITY INDEX (MODI) | 3rd week
  ODI is a reliable and valid to assess the functional disability related to low back pain,
  it has 10 questions, each question is answered via six choices, the first statement takes 0 and the sixth statement take 5, the patient was asked to selected the best chouce that prescribe her disability, then all scores collected and taken as a percentage from the total score the higher score indicate great disability, scores from 0-20% denote minimal disability, scores 40-60% denote moderate disability, while scores from 60-80% denote crippled disability , finally scores from 80-100% represent patient who are confined to bed. Changes from the baseline and 3rd week.

SECONDARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 3rd week
  Changes from baseline the Numeric Pain Rating Scale (NPRS) is a unidimensional measure of pain intensity in adults. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable"). Changes from the baseline and 3rd week.

CONTACTS AND LOCATIONS:
Overall Officials: Afifa Safdar, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Syed Medical Complex., Sialkot, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ostgaard HC, Andersson GB, Wennergren M. The impact of low back and pelvic pain in pregnancy on the pregnancy outcome. Acta Obstet Gynecol Scand. 1991;70(1):21-4. doi: 10.3109/00016349109006172. PMID 1830444
- [Background] To WW, Wong MW. Factors associated with back pain symptoms in pregnancy and the persistence of pain 2 years after pregnancy. Acta Obstet Gynecol Scand. 2003 Dec;82(12):1086-91. doi: 10.1046/j.1600-0412.2003.00235.x. PMID 14616251
- [Background] Berg G, Hammar M, Moller-Nielsen J, Linden U, Thorblad J. Low back pain during pregnancy. Obstet Gynecol. 1988 Jan;71(1):71-5. PMID 2962023
- [Background] Hayden JA, Ellis J, Ogilvie R, Malmivaara A, van Tulder MW. Exercise therapy for chronic low back pain. Cochrane Database Syst Rev. 2021 Sep 28;9(9):CD009790. doi: 10.1002/14651858.CD009790.pub2. PMID 34580864
- [Background] Puntumetakul R, Saiklang P, Tapanya W, Chatprem T, Kanpittaya J, Arayawichanon P, Boucaut R. The Effects of Core Stabilization Exercise with the Abdominal Drawing-in Maneuver Technique versus General Strengthening Exercise on Lumbar Segmental Motion in Patients with Clinical Lumbar Instability: A Randomized Controlled Trial with 12-Month Follow-Up. Int J Environ Res Public Health. 2021 Jul 23;18(15):7811. doi: 10.3390/ijerph18157811. PMID 34360103
- [Background] Javadov A, Ketenci A, Aksoy C. The Efficiency of Manual Therapy and Sacroiliac and Lumbar Exercises in Patients with Sacroiliac Joint Dysfunction Syndrome. Pain Physician. 2021 May;24(3):223-233. PMID 33988941